CLINICAL TRIAL: NCT05315791
Title: Clinical Application Strategies of Maxillary Sinus Buccal Bony Window With Different Residual Bone Heights in Lateral Maxillary Sinus Floor Elevation
Brief Title: Clinical Application Strategies of Maxillary Sinus Buccal Bony Window
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Guoli Yang, Director, The Dental Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-126
Record Dates: First submitted 2022-03-12; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Sinus Floor Augmentation; Maxillary Sinus
Keywords: maxillary sinus floor elevation; CBCT; RCT

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- a: ground into pieces (Experimental): 0~3mm
  Interventions: Procedure: different methods for maxillary sinus floor elevation
- b: replace the bone (Experimental): 0~3mm
  Interventions: Procedure: different methods for maxillary sinus floor elevation
- c: turn inward (Experimental): 0~3mm
  Interventions: Procedure: different methods for maxillary sinus floor elevation
- d: ground into pieces (Experimental): 3~5mm
  Interventions: Procedure: different methods for maxillary sinus floor elevation
- e: replace the bone (Experimental): 3~5mm
  Interventions: Procedure: different methods for maxillary sinus floor elevation
- f: turn inward (Experimental): 3~5mm
  Interventions: Procedure: different methods for maxillary sinus floor elevation

INTERVENTIONS:
Procedure: different methods for maxillary sinus floor elevation — a: 0~3mm+ground into pieces; b: 0~3mm+replace the bone; c: 0~3mm+turn inward to hold up the membrane; d: 3~5mm+ground into pieces; e: 3~5mm+replace the bone; f: 3~5mm+turn inward to hold up the membrane

SUMMARY:
Through randomized controlled trials, investigators will recruit participants who need maxillary sinus floor elevation with different residual bone height, and utilize the maxillary sinus buccal bony window during the surgery. Then investigators will gather the related information of participants, collect and analyze their CBCT data, in order to help surgeons select the best operating method for different patients.

DETAILED DESCRIPTION:
Through randomized controlled trials, investigators will recruit 60 participants who need maxillary sinus floor elevation with different residual bone height (0~3mm; 3~5mm), and utilize the maxillary sinus buccal bony window during the surgery (A: ground into pieces; B: replace the bone; C: turn inward to hold up the membrane). Then investigators will gather the related information of participants, collect and analyze their CBCT data, in order to help surgeons select the best operating method for different patients.

ELIGIBILITY:
Inclusion Criteria:

* A single maxillary posterior tooth was missing, and the missing time was ≥ 3 months
* Gingival distance ≥ 4mm
* Residual bone height ≤ 5mm and residual bone width ≥ 6mm
* Good systemic health
* CBCT image was complete and clear, and there was no obvious artifact affecting the measurement
* Informed consent.

Exclusion Criteria:

* Untreated diabetes or other serious systemic diseases
* Untreated periodontal disease
* Uncontrolled periapical lesions of adjacent teeth
* Certain bone diseases such as osteoporosis and osteosclerosis
* Severe night bruxism
* Mental illness
* Pregnant or breast-feeding patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-03-02 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
ABH change | baseline, 6 months, and 1, 2, 3, 5, 10 years after the surgery
  Apical bone height (ABH): Represented the grafted height at baseline and the grafted height with neo-formed bone at follow-ups.
ESBG change | baseline, 6 months, and 1, 2, 3, 5, 10 years after the surgery
  Endo-sinus bone gain (ESBG): ESBG = ABH + implant protrusion length at baseline; ESBG represented the grafted height and neo-formed bone, and described the height difference of radiopaque area in the sinus cavity at different times.
RBH | baseline
  Residual bone height (RBH): Only assessed at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Stomatology, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Starch-Jensen T, Jensen JD. Maxillary Sinus Floor Augmentation: a Review of Selected Treatment Modalities. J Oral Maxillofac Res. 2017 Sep 30;8(3):e3. doi: 10.5037/jomr.2017.8303. eCollection 2017 Jul-Sep. PMID 29142655
- [Result] Niu L, Wang J, Yu H, Qiu L. New classification of maxillary sinus contours and its relation to sinus floor elevation surgery. Clin Implant Dent Relat Res. 2018 Aug;20(4):493-500. doi: 10.1111/cid.12606. Epub 2018 Apr 25. PMID 29691967
- [Result] Zhou Y, Shi Y, Si M, Wu M, Xie Z. The comparative evaluation of transcrestal and lateral sinus floor elevation in sites with residual bone height </=6 mm: A two-year prospective randomized study. Clin Oral Implants Res. 2021 Feb;32(2):180-191. doi: 10.1111/clr.13688. Epub 2020 Dec 26. PMID 33220090